CLINICAL TRIAL: NCT07269808
Title: Sedation During Endoscopy Using Remimazolam: Efficacy in a Novel Exploration (SERENE)
Brief Title: Sedation During Endoscopy Using Remimazolam: Efficacy in a Novel Exploration
Acronym: SERENE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Chair, Department of Anesthesiology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025P002893
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Sedation; Endoscopy
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm Title: Remimazolam Sedation (Experimental): Participants randomized to this arm will receive remimazolam 0.20 mg/kg for procedural sedation. The maximum initial bolus will be 15 mg, with additional doses administered in 2.5 mg increments as needed to maintain adequate sedation. Intravenous fentanyl (25-100 mcg) may be administered as an adjunct per clinician judgement. This dosing strategy reflects the institution's standard-of-care approach to remimazolam-based sedation.
  Interventions: Drug: Remimazolam
- Propofol Sedation (Active Comparator): Participants randomized to this arm will receive propofol up to 1.5 mg/kg as the initial bolus, followed by intermittent boluses of 10-40 mg according to routine clinical practice. Intravenous fentanyl (25-100 mcg) may be administered as an adjunct per clinician judgement. This regimen reflects the institution's standard-of-care approach to propofol-based sedation.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam will be administered at 0.20 mg/kg for procedural sedation. The maximum initial bolus is 15 mg, with additional 2.5 mg doses given as needed to maintain sedation. Intravenous fentanyl (25-100 mcg) may be used adjunctively per clinician judgement
  Other Names: Byfavo
  Arms: Arm Title: Remimazolam Sedation
Drug: Propofol — Propofol will be administered with an initial bolus of up to 1.5 mg/kg, followed by intermittent 10-40 mg boluses according to routine clinical practice. Intravenous fentanyl (25-100 mcg) may be used adjunctively per clinician judgement.
  Other Names: Diprivan
  Arms: Propofol Sedation

SUMMARY:
This study is a pragmatic, randomized controlled pilot trial comparing remimazolam with propofol for endoscopic procedures, designed to assess the feasibility and clinical outcomes associated with implementing a pragmatic randomized trial of sedation practices in the endoscopy setting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age or older
* Planned endoscopic procedure
* American Society of Anesthesiologists (ASA) Physical Status I to III

Exclusion Criteria:

* Planned tracheal intubation
* Procedure length anticipated to exceed 45 minutes
* Previously participated in the trial
* Pregnant (defined as a positive test using pre-procedural clinical testing performed as part of their routine care) or breastfeeding
* Allergy or hypersensitivity to one of the study medications
* Blind, deaf, or unable to communicate in English
* Co-enrollment in other interventional studies that, in the opinion of the site investigator and/or their delegate, might interfere with study participation, collection, or interpretation of the study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Meeting Inclusion/Exclusion Criteria | From initiation of screening through end of study enrollment period.
  Counts the number of patients screened who meet all prespecified inclusion and exclusion criteria for trial eligibility.
Number of Patients Consented | From initiation of recruitment through end of study enrollment period.
  Total number of eligible patients who provide informed consent to participate in the study.
Number of Patients Receiving the Randomized Intervention Per Protocol | From randomization through completion of the endoscopic procedure.
  Number of consented participants who are successfully randomized and receive their assigned sedation intervention according to the study protocol without major deviations.
Number of Completed Questionnaires | At the end of the procedure and at the immediate post-procedure assessment.
  Total number of study-related questionnaires completed by participants at the designated assessment time points, used to evaluate feasibility and acceptability of study procedures.

OTHER OUTCOMES:
Incidence and Duration of Adverse Clinical Events | From induction of sedation through end of the procedure
  Incidence and duration of predefined adverse clinical events, including respiratory insufficiency, hypoxemia, hypotension, and bradycardia, occurring during the procedure.
Procedural Success | From induction of sedation through end of the procedure
  Proportion of procedures completed successfully, defined as full completion of the planned endoscopic procedure with the patient maintaining adequate spontaneous ventilation throughout.
Patient Satisfaction | At the immediate post-procedure assessment
  Patient-reported satisfaction with the procedural sedation experience, assessed using a standardized post-procedure satisfaction questionnaire.
Provider Satisfaction | Immediately after procedure completion
  Satisfaction ratings from nurses, endoscopists, and anesthesiologists regarding the sedation process, collected using standardized provider questionnaire instruments.
Procedure Duration | From the start of the procedure through the end of the procedure
  Total time from procedure start (scope insertion) to procedure end (scope removal), recorded in minutes.
Post Anesthesia Care Unit Length of Stay | Perioperative/Periprocedural
  Time from the end of the endoscopic procedure to achievement of standardized post-anesthesia care unit discharge criteria.
Time From Induction of Sedation to Procedure Start | From induction of sedation to procedure start
  Interval between administration of the initial sedation dose and the start of the endoscopic procedure (scope insertion).
Richmond Agitation-Sedation Scale (RASS) Scores | Repeated measures assessed from induction of sedation through end of the procedure
  Sedation depth assessed using repeated RASS measurements at prespecified intervals throughout the procedure.
Oxygen Saturation | Repeated measures assessed from induction of sedation through end of the procedure
  Continuous or intermittent oxygen saturation (SpO₂) measurements collected at prespecified intervals during the procedure.
Blood Pressure Measurements | Repeated measures assessed from induction of sedation through end of the procedure
  Repeated assessments of systolic, diastolic, and mean arterial blood pressure at prespecified intervals during the procedure.
Unplanned Conversion to General Anesthesia or Use of Non-Study Sedative | From sedation induction through end of procedure.
  Number of cases requiring conversion to general anesthesia or administration of any sedative agent outside the assigned study drug protocol
Total Fentanyl Dose Administered | From induction of sedation to procedure end
  Cumulative dose of intravenous fentanyl administered as an adjunct to sedation during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwaseun Johnson-Akeju, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol